CLINICAL TRIAL: NCT00285688
Title: Antibiotic Resistance Helicobacter Pylori and Clarithromycin Resistance Mutation in Helicobacter Pylori in Rajavithi Hospital
Brief Title: Antibiotic Resistant Helicobacter Pylori in Rajavithi Hospital
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Dr Piyathida Harnsomburana, Biomolecular Research Center, Rajavithi hospital: Thailand
Other Study IDs: RH-CMR-002
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dyspepsia
Keywords: H. Pylori, Clarithromycin resistant, gene
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric Biopsy tissue and H. pylori DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Gastroscope positive for H. pylori and resistant to clarithromycin
  Interventions: Procedure: gastroscopic examination
- 2: Gastroscope positive for H. pylori and not resistant to clarithromycin
  Interventions: Procedure: gastroscopic examination

INTERVENTIONS:
Procedure: gastroscopic examination — gastroscopic examination for tissue biopsy and real time PCR for gene study

SUMMARY:
Peptic ulcer disease is the most common gastrointestinal disease. Antibiotic resistant Helicobacter pylori is a major problem worldwide. The gold standard for Helicobacter pylori eradication is composed of Proton-pump inhibitor/Ranitidine bismuth citrate + Amoxycillin + Metronidazole /Clarithromycin. In Thailand, clarithromycin resistant strains increased and led to treatment failure. Data on file at Rajavithi Hospital showed that metronidazole resistant H. pylori was about 50% and Clarithromycin resistant strains accounted for 8%. This molecular genetic study will be performed in patients presenting with dyspepsia, who had an indication for gastroscopic examination, to explore the incidence of antibiotic resistant Helicobacter pylori in Rajavithi Hospital, Thailand.

DETAILED DESCRIPTION:
Genetic and Biomolecular factors determining clarithromycin resistance will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* male or female with dyspepsia
* age > 15 years
* fulfil indication for gastroscopic examination
* able to give informed consent

Exclusion Criteria:

* contraindication for gastroscopic examination and biopsy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dydpepsia patient with gastroscopic examination
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-06 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of H. pylori Clarithromycin resistance gene | one year

SECONDARY OUTCOMES:
Characteristic of H. pylori clarithromycin resistant gene mutation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Piyathida Harnsoomboon, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Derived] Hansomburana P, Anantapanpong S, Sirinthornpunya S, Chuengyong K, Rojborwonwittaya J. Prevalence of single nucleotide mutation in clarithromycin resistant gene of Helicobacter pylori: a 32-months prospective study by using hybridization real time polymerase chain reaction. J Med Assoc Thai. 2012 Mar;95 Suppl 3:S28-35. PMID 22619884